CLINICAL TRIAL: NCT04203160
Title: A Multi-Center Randomized Phase IB/II Study of Gemcitabine and Cisplatin With or Without CPI-613 as First Line Therapy for Patients With Advanced Unresectable Biliary Tract Cancer (BilT-04)
Brief Title: Gemcitabine and Cisplatin With or Without CPI-613 as First Line Therapy for Patients With Advanced Unresectable Biliary Tract Cancer (BilT-04)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2019.116; HUM00170490 (Other: University of Michigan)
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Cancer
Keywords: Cholangiocarcinoma; Gallbladder cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — devimistat; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: Phase II: 2:1 Randomization with Bayesian Design Control Arm
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 and Phase 2, Arm A (investigational) (Experimental): On Day 1 and Day 8 of each 3-week cycle, patients will receive CPI-613 + gemcitabine and cisplatin. Patients may continue gemcitabine, cisplatin and CPI-613 for up to 2 years in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: CPI 613; Drug: Gemcitabine; Drug: Cisplatin
- Phase 2, Arm B (standard of care) (Active Comparator): On Day 1 and Day 8 of each 3-week cycle, patients will receive gemcitabine and cisplatin. Patients may continue gemcitabine and cisplatin for up to 2 years in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: CPI 613 — Given intravenously
  Other Names: Devimistat®
  Arms: Phase 1 and Phase 2, Arm A (investigational)
Drug: Gemcitabine — Given intravenously
  Other Names: Gemzar®
Drug: Cisplatin — Given intravenously
  Other Names: CDDP, Platinol®, NSC-119875

SUMMARY:
The purpose of this research study is to determine the safety and efficacy of CPI-613 (devimistat) in the treatment of advanced biliary tract cancer when used in combination with standard of care chemotherapy (gemcitabine plus cisplatin) compared to gemcitabine plus cisplatin alone.

This research study has two parts:

In the phase 1 portion of this study, patients will receive a combination of CPI-613 and standard of care chemotherapy. Dose levels of CPI-613 will be adjusted to find the best dose, which will be the recommended phase 2 dose level.

In the phase 2 portion of this study, patients will be randomized into two arms. Patients in Arm A will receive the combination of the recommended dose level of CPI-613 and standard of care chemotherapy. Patients in Arm B will receive standard of care chemotherapy.

At the end of the study, researchers will compare the health outcomes of the patients that received CPI-613 + standard care to the outcomes of patients that received only standard care.

ELIGIBILITY:
Inclusion:

* Patients must have a pathologically or cytologically confirmed carcinoma (except neuroendocrine) of the biliary tract (intra-hepatic, extra-hepatic (hilar, distal) or gallbladder) that is not eligible for curative resection, transplantation, or ablative therapies. Tumors of mixed cholangiocarcinoma/hepatocellular carcinoma histology are excluded.
* Patients may not have received prior systemic treatment (chemotherapy or targeted therapy) for advanced BTC. Prior peri-operative chemotherapy is permitted provided it was completed > 6 months from enrollment.
* Patients may have received prior radiation, chemoembolization, radioembolization or other local ablative therapies or hepatic resection if completed ≥ 4 weeks prior to enrollment AND if patient has recovered to ≤ grade 1 toxicity. Extrahepatic palliative radiation is permitted if completed ≥ 2 weeks prior to enrollment AND if patient has recovered to ≤ grade 1 toxicity
* Patients must have radiographically measurable disease (as per RECISTv1.1) in at least one site not previously treated with radiation or liver directed therapy (including bland, chemo- or radio-embolization, or ablation) either within the liver or in a metastatic site.
* Must be ≥ 18 years of age.
* Must have an ECOG performance status of 0-1.
* Ability to understand and willingness to sign IRB-approved informed consent.
* Willing to provide archived tissue, if available, from a previous diagnostic biopsy or surgery.
* Must be able to tolerate CT and/or MRI with contrast.
* Adequate organ function (per protocol) obtained ≤ 2 weeks prior to enrollment.
* Women of child-bearing potential and men must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) OR abstinence prior to study entry, for the duration of study participation and for 6 months (for men and women) following completion of study therapy.

Exclusions:

* Prior history of brain metastasis (unless previously treated, asymptomatic and stable for at least 3 months) or organ transplant.
* Underwent a major surgical procedure < 4 weeks prior to enrollment.
* Active second malignancy other than in situ cancer or localized prostate cancer (Gleason score <8). Patients with history of other malignancy are eligible provided primary treatment of that cancer was completed > 1 year prior to enrollment and the patient is free of clinical or radiologic evidence of recurrent or progressive malignancy.
* Ongoing active, uncontrolled infection (must be afebrile for > 48 hours off antibiotics) .
* Psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements.
* Pregnancy or breastfeeding. (Women must not be pregnant or breastfeeding since study drugs may harm the fetus or child. All females of childbearing potential [not surgically sterilized and between menarche and 1 year post menopause] must have a negative screening pregnancy test.)
* Active heart disease including symptomatic heart failure (NYHA class 3 or 4), unstable angina pectoris, uncontrolled cardiac arrhythmia or interstitial lung disease.
* Prisoners or subjects who are involuntarily incarcerated, or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness would be excluded.
* Prolonged QTcF interval >480 msec.
* Known hypersensitivity to cisplatin, gemcitabine or CPI-613, or its inactive components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Sahai, MBBS, MS, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (10):
- United States (10):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Northwestern University -- Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Atlantic Health System, Morristown, New Jersey
  - University Hospitals - Seidman Cancer Center, Cleveland, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern -- Simmons Comprehensive Cancer Center, Dallas, Texas
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2, Arm A (Investigational); Phase 1, CPI-613 500 mg/m2; Phase 1, CPI-613 1000 mg/m2; Phase 1, CPI-613 1500 mg/m2; Phase 1, CPI-613 2000 mg/m2: On Day 1 and Day 8 of each 3-week cycle, patients will receive CPI-613 + gemcitabine and cisplatin. Patients may continue gemcitabine, cisplatin and CPI-613 for up to 2 years in absence of disease progression or unacceptable toxicity.
  CPI 613: Given intravenously
  Gemcitabine: Given intravenously
  Cisplatin: Given intravenously
Period: Overall Study
Arm/Group | Phase 2, Arm A (Investigational) | Phase 2, Arm B (Standard of Care) | Phase 1, CPI-613 500 mg/m2 | Phase 1, CPI-613 1000 mg/m2 | Phase 1, CPI-613 1500 mg/m2 | Phase 1, CPI-613 2000 mg/m2
Started | 37 | 18 | 1 | 1 | 2 | 16
Completed | 19 | 6 | 0 | 1 | 2 | 10
Not Completed | 18 | 12 | 1 | 0 | 0 | 6
Not completed — Alternative Therapy | 3 | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 5 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 7 | 5 | 0 | 0 | 0 | 0
Not completed — Sponsor Termination | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1, CPI-613 500 mg/m2: On Day 1 and Day 8 of each 3-week cycle, patients will receive CPI-613 + gemcitabine and cisplatin. Patients may continue gemcitabine, cisplatin and CPI-613 for up to 2 years in absence of disease progression or unacceptable toxicity.
  CPI 613: Given intravenously
  Gemcitabine: Given intravenously
- Total: Total of all reporting groups
Arm/Group | Phase 2, Arm A (Investigational) | Phase 2, Arm B (Standard of Care) | Phase 1, CPI-613 500 mg/m2 | Phase 1, CPI-613 1000 mg/m2 | Phase 1, CPI-613 1500 mg/m2 | Phase 1, CPI-613 2000 mg/m2 | Total
Number analyzed (Participants) | 37 | 18 | 1 | 1 | 2 | 16 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 4 | 0 | 0 | 2 | 6 | 25
  >=65 years | 24 | 14 | 1 | 1 | 0 | 10 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 1 | 0 | 2 | 6 | 37
  Male | 21 | 6 | 0 | 1 | 0 | 10 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 0 | 0 | 1 | 1 | 10
  Not Hispanic or Latino | 32 | 15 | 1 | 1 | 1 | 14 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 34 | 15 | 1 | 1 | 2 | 13 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 37 | 18 | 1 | 1 | 2 | 16 | 75

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Incidence of Dose-limiting Toxicity
Description: Dose limiting toxicities will determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of combination therapy with CPI-613 + gemcitabine and cisplatin. Assessed using the NCI CTCAE v5.0
Time Frame: Up to day 22
Population: only applies to Phase 1 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Arm A (Investigational) | Phase 2, Arm B (Standard of Care) | Phase 1, CPI-613 500 mg/m2 | Phase 1, CPI-613 1000 mg/m2 | Phase 1, CPI-613 1500 mg/m2 | Phase 1, CPI-613 2000 mg/m2
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 2 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: Objective response assessment will be determined by review of CT or MR scans of the chest, abdomen and pelvis. ORR (Partial Response + Complete Response) will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, during active study treatment. All enrolled patients who receive at least 1 cycle of therapy and have their disease re-evaluated will be considered evaluable for response. (Note: Patients who exhibit objective disease progression prior to the end of cycle 1 will also be considered evaluable.)
Time Frame: Until last dose of study treatment (up to 2 years)
Population: Phase 2, Arm A- 37 patients were randomized to Arm A treatment, with 36 patients receiving treatment. Per protocol the 16 patients in the Phase 1 portion of the study were included, for a total of 52 patients in the investigational arm. All 52 subjects were considered for evaluability. Two subjects were found to be unevaluable.
  Phase 2, Arm B- 18 patients were randomized to Arm B treatment, with 16 patients receiving treatment.Three subjects were found to be unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Arm A (Investigational) | Phase 2, Arm B (Standard of Care) | Phase 1, CPI-613 500 mg/m2 | Phase 1, CPI-613 1000 mg/m2 | Phase 1, CPI-613 1500 mg/m2 | Phase 1, CPI-613 2000 mg/m2
Number analyzed (Participants) | 50 | 13 | 0 | 0 | 0 | 0
Participants | 15 | 6 | 0 | 0 | 0 | 0

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS will be determined from date of first study treatment until the date of radiological or clinical progression (leading to withdrawal from the study) or date of last disease evaluation (for patients without progression). It will be calculated using the product-limit method of Kaplan and Meier. All patients that receive at least one dose of study treatment will be considered evaluable.
Time Frame: Until last dose of study treatment (up to 2 years)
Population: Phase 2, Arm A- 37 patients were randomized to Arm A treatment, with 36 patients receiving treatment. Per protocol the 16 patients in the Phase 1 portion of the study were included, for a total of 52 patients in the investigational arm. All 52 subjects were considered for evaluability. Two subjects were found to be unevaluable.
  Phase 2, Arm B- 18 patients were randomized to Arm B treatment, with 16 patients receiving treatment. Three subjects were found to be unevaluable.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Arm A (Investigational) | Phase 2, Arm B (Standard of Care) | Phase 1, CPI-613 500 mg/m2 | Phase 1, CPI-613 1000 mg/m2 | Phase 1, CPI-613 1500 mg/m2 | Phase 1, CPI-613 2000 mg/m2
Number analyzed (Participants) | 50 | 13 | 0 | 0 | 0 | 0
months | 8.7 [5.8 to 11.3] | 9.6 [7.3 to NA] — not yet estimable as trial was terminated by the sponsor |  |  |  |

4. Secondary Outcome: Median Overall Survival (OS)
Description: From date of first study treatment until date of last disease evaluation or until death from any cause. Using the product-limit method of Kaplan and Meier.
Time Frame: Up to 3 years after enrollment
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Arm A (Investigational) | Phase 2, Arm B (Standard of Care) | Phase 1, CPI-613 500 mg/m2 | Phase 1, CPI-613 1000 mg/m2 | Phase 1, CPI-613 1500 mg/m2 | Phase 1, CPI-613 2000 mg/m2
Number analyzed (Participants) | 50 | 13 | 0 | 0 | 0 | 0
months | 15.6 [11.8 to 22.5] | 22.2 [8.6 to NA] — NA as not yet estimable as trial was terminated by the sponsor |  |  |  |

5. Secondary Outcome: Incidence of Toxicities
Description: To evaluate the safety of CPI-613 in combination with gemcitabine and cisplatin in this patient population, assessed using the Common Toxicity Criteria for Adverse Events (CTCAE) v5.0. All patients that receive at least one dose of study treatment will be considered evaluable. Number of patients experiencing the maximum graded toxicity (Grade 2 or higher).
Time Frame: Up to 100 days after last dose of study treatment
Population: Phase 2, Arm A- 37 patients were randomized to Arm A treatment, with 36 patients receiving treatment. Per protocol the 16 patients receiving the RP2D of Devimistat in the Phase 1 portion of the study were included, for a total of 52 patients. This combination was done per protocol.
  Phase 2, Arm B- 18 patients were randomized to Arm B treatment, with 16 patients receiving treatment. For 16 receiving study treatment
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1, Arm A (Investigational); Phase 2, Arm A (Investigational): On Day 1 and Day 8 of each 3-week cycle, patients will receive CPI-613 + gemcitabine and cisplatin. Patients may continue gemcitabine, cisplatin and CPI-613 for up to 2 years in absence of disease progression or unacceptable toxicity.
  CPI 613: Given intravenously
  Gemcitabine: Given intravenously
  Cisplatin: Given intravenously
Arm/Group | Phase 1, Arm A (Investigational) | Phase 2, Arm A (Investigational) | Phase 2, Arm B (Standard of Care)
Number analyzed (Participants) | 0 | 52 | 16
Participants
  Abdominal pain- Grade 3 |  | 1 | 0
  Alanine aminotransferase increased- Grade 2 |  | 1 | 0
  Alopecia- Grade 2 |  | 2 | 1
  Anemia- Grade 2 |  | 4 | 2
  Anemia- Grade 3 |  | 10 | 7
  Anorexia- Grade 2 |  | 3 | 4
  Anorexia- Grade 3 |  | 1 | 0
  Aspartate aminotransferase increased- Grade 2 |  | 1 | 0
  Bacteremia- Grade 2 |  | 1 | 0
  Biliary tract Infection- Grade 2 |  | 1 | 0
  Blood transfusion- Grade 2 |  | 1 | 0
  Blood bilirubin increased- Grade 2 |  | 1 | 0
  chest tightness- Grade 2 |  | 1 | 0
  Cholecystitis- Grade 3 |  | 1 | 0
  Constipation- Grade 2 |  | 3 | 0
  Creatinine increased- Grade 2 |  | 3 | 1
  Diarrhea- Grade 2 |  | 1 | 0
  Diarrhea- Grade 3 |  | 1 | 1
  Dysgeusia- Grade 2 |  | 2 | 0
  Enterocolitis- Grade 3 |  | 1 | 0
  Fatigue- Grade 2 |  | 15 | 3
  Fatigue- Grade 3 |  | 3 | 0
  Febrile Neutropenia- Grade 3 |  | 1 | 0
  Flu like symptoms- Grade 2 |  | 1 | 0
  Gastroesophageal relux disease- Grade 2 |  | 1 | 1
  hypersalivation- Grade 2 |  | 1 | 0
  generalize muscle weakness- Grade 2 |  | 1 | 0
  Hematuria- Grade 3 |  | 1 | 0
  Hiccups- Grade 2 |  | 1 | 1
  Hot flashes- Grade 2 |  | 1 | 0
  Hypercalcemia- Grade 3 |  | 1 | 0
  Hyperglycemia- Grade 2 |  | 2 | 0
  Hypertension- Grade 2 |  | 1 | 0
  Hypertension- Grade 3 |  | 1 | 0
  Hypoalbuminemia- Grade 2 |  | 1 | 0
  Hypokalemia- Grade 2 |  | 3 | 1
  Hypomagnesemia- Grade 2 |  | 3 | 1
  Hypomagnesemia- Grade 3 |  | 1 | 0
  Hyponatremia- Grade 3 |  | 2 | 0
  Infection- Grade 3 |  | 1 | 0
  Infusion Related Reaction- Grade 2 |  | 3 | 1
  Lymphocyte count decreased- Grade 3 |  | 1 | 1
  Nausea- Grade 2 |  | 8 | 2
  Neutrophil count decreased- Grade 2 |  | 2 | 1
  Neutrophil count decreased- Grade 3 |  | 18 | 8
  Neutrophil count decreased- Grade 4 |  | 2 | 0
  Pancreatitis- Grade 3 |  | 1 | 0
  Peripheral Motor Neuropathy- Grade 2 |  | 1 | 0
  Peripheral Sensory Neuropathy- Grade 2 |  | 3 | 0
  Platelet count decreased- Grade 2 |  | 3 | 2
  Platelet count decreased- Grade 3 |  | 5 | 0
  Platelet count decreased- Grade 4 |  | 2 | 1
  Sepsis- Grade 3 |  | 1 | 0
  Stroke- Grade 3 |  | 1 | 0
  Pulmonary Embolism- Grade 3 |  | 1 | 0
  Urinary Tract Infection- Grade 2 |  | 1 | 0
  Vomiting- Grade 2 |  | 2 | 1
  White Blood Cell Decreased- Grade 2 |  | 3 | 0
  White Blood Cell Decreased- Grade 3 |  | 4 | 1
  Alanine aminotransferase increased- Grade 3 |  | 0 | 1
  Aspartate aminotransferase increased- Grade 3 |  | 0 | 1
  Fever- Grade 2 |  | 0 | 1
  Generalized Edema- Grade 2 |  | 0 | 1
  Liver Abscess- Grade 3 |  | 0 | 1
  Hypomagnesemia- Grade 4 |  | 0 | 1
  Lymphocyte count decreased- Grade 4 |  | 0 | 1

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment. Up to 2 years. All-Cause Mortality monitored/assessed up to 3 years
Arm/Group | Phase 2, Arm A (Investigational) | Phase 2, Arm B (Standard of Care) | Phase 1, CPI-613 500 mg/m2 | Phase 1, CPI-613 1000 mg/m2 | Phase 1, CPI-613 1500 mg/m2 | Phase 1, CPI-613 2000 mg/m2
All-Cause Mortality (participants affected / at risk) | 25/37 | 7/18 | 0/1 | 1/1 | 2/2 | 12/16
Serious Adverse Events (participants affected / at risk) | 13/37 | 9/18 | 0/1 | 1/1 | 2/2 | 11/16
Other Adverse Events (participants affected / at risk) | 35/37 | 15/18 | 1/1 | 1/1 | 2/2 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2, Arm A (Investigational) (N=37) | Phase 2, Arm B (Standard of Care) (N=18) | Phase 1, CPI-613 500 mg/m2 (N=1) | Phase 1, CPI-613 1000 mg/m2 (N=1) | Phase 1, CPI-613 1500 mg/m2 (N=2) | Phase 1, CPI-613 2000 mg/m2 (N=16)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fever (General disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (7) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Progressive Disease (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
biliary obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Giardiasis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2, Arm A (Investigational) (N=37) | Phase 2, Arm B (Standard of Care) (N=18) | Phase 1, CPI-613 500 mg/m2 (N=1) | Phase 1, CPI-613 1000 mg/m2 (N=1) | Phase 1, CPI-613 1500 mg/m2 (N=2) | Phase 1, CPI-613 2000 mg/m2 (N=16)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (20) | 6 (7) | 0 (0) | 1 (1) | 2 (5) | 9 (17)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 3 (9)
Alkaline phosphatase increased (Investigations) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
Allergic reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (General disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Anemia (Investigations) | 12 (58) | 11 (25) | 1 (2) | 0 (0) | 2 (15) | 8 (24)
Anorexia (General disorders) | 9 (9) | 7 (7) | 0 (0) | 1 (5) | 2 (5) | 5 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 4 (7) | 2 (5) | 0 (0) | 0 (0) | 1 (6) | 3 (6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (General disorders) | 5 (5) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Bloating (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 5 (9)
Blurred vision (Eye disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Bone pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (17) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 9 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (11)
Cystitis noninfective (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (9) | 4 (6) | 0 (0) | 1 (1) | 1 (2) | 10 (18)
Dizziness (General disorders) | 8 (8) | 6 (9) | 0 (0) | 1 (1) | 0 (0) | 3 (7)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 6 (8) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Dyspepsia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysphagia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 5 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Enterocolitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Epistaxis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 25 (44) | 8 (12) | 0 (0) | 1 (3) | 2 (3) | 15 (24)
Febrile neutropenia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fever (General disorders) | 3 (5) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 4 (6)
Flank pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric hemorrhage (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Generalized edema (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Generalized muscle weakness (General disorders) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatic infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hoarseness (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Investigations) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Hyperhidrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (2) | 1 (1) | 0 (0) | 1 (3) | 4 (8)
Hyperuricemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Investigations) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypokalemia (Investigations) | 5 (11) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Investigations) | 9 (21) | 4 (21) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Investigations) | 3 (5) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Infections and infestations) | 5 (8) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (6) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (General disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscle cramp (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness lower limb (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (24) | 6 (8) | 1 (1) | 1 (3) | 2 (2) | 11 (16)
Neck pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 15 (33) | 10 (17) | 1 (3) | 1 (5) | 1 (10) | 10 (19)
Oral dysesthesia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (General disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Peritoneal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 10 (27) | 5 (8) | 0 (0) | 0 (0) | 1 (8) | 5 (22)
Pleural effusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 6 (7) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Thrush (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attacks (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (16) | 3 (3) | 0 (0) | 1 (2) | 1 (2) | 6 (11)
Weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 5 (16) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT04203160/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT04203160/ICF_001.pdf